CLINICAL TRIAL: NCT03081234
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of Ribociclib With Endocrine Therapy as an Adjuvant Treatment in Patients With Hormone Receptor-positive, HER2-negative, Intermediate Risk Early Breast Cancer
Brief Title: Adjuvant Ribociclib With Endocrine Therapy in Hormone Receptor+/HER2- Intermediate Risk Early Breast Cancer
Acronym: EarLEE-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn due to change in plan for this study and not due to safety reasons.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLEE011H2301
Record Dates: First submitted 2017-03-01; First posted 2017-03-16 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Hormone receptor-positive; Estrogen and/or progesterone receptor-positive; HER2-negative; Intermediate risk early breast cancer; Adjuvant; Ribociclib; LEE011; CDK4/6 inhibitor; Endocrine therapy; Phase III; breast carcinoma; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib + adjuvant endocrine therapy (Experimental): Ribociclib in combination with standard adjuvant endocrine therapy
  Interventions: Drug: Ribociclib; Drug: Adjuvant endocrine therapy
- Placebo + adjuvant endocrine therapy (Active Comparator): Placebo in combination with standard adjuvant endocrine therapy
  Interventions: Drug: Placebo; Drug: Adjuvant endocrine therapy

INTERVENTIONS:
Drug: Ribociclib — Ribociclib 600 mg daily on days 1 to 21 of a 28-day cycle for 26 cycles (approximately 24 months). Ribociclib will be supplied in the form of 200 mg tablets.
  Other Names: LEE011
  Arms: Ribociclib + adjuvant endocrine therapy
Drug: Placebo — Placebo 600 mg daily on days 1 to 21 of a 28-day cycle for 26 cycles (approximately 24 months). Placebo will be supplied in the form of 200 mg tablets.
  Arms: Placebo + adjuvant endocrine therapy
Drug: Adjuvant endocrine therapy — Tamoxifen 20 mg daily, or letrozole 2.5 mg daily, or anastrozole 1 mg daily, or exemestane 25 mg daily (male patients will be treated with tamoxifen 20 mg daily) for a total duration of at least 60 months. In premenopausal women, adjuvant endocrine therapy may include GnRH agonist administered every 28 days.

SUMMARY:
This is an international, multi-center, randomized, double-blinded, placebo-controlled clinical study evaluating the efficacy and safety of ribociclib with endocrine therapy as an adjuvant treatment in patients with hormone receptor-positive, HER2-negative, intermediate risk breast cancer.

DETAILED DESCRIPTION:
While adjuvant endocrine therapy (ET) is effective in reducing risk of recurrence in patients with hormone receptor (HR)-positive early breast cancer (EBC), recurrences are still common, especially in patients with unfavorable clinical, pathological and/or molecular features. Ribociclib, a CDK4/6 inhibitor, demonstrated clinical efficacy with tolerable toxicity when added to ET in patients with HR-positive, HER2-negative advanced breast cancer. The purpose of this study is to evaluate the effect of addition of ribociclib to standard adjuvant ET on invasive disease-free survival in patients with HR+, HER2- intermediate-risk EBC.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed unilateral primary invasive adenocarcinoma of the breast
* Estrogen receptor-positive and/or progesterone receptor-positive, HER2-negative breast cancer
* Patient is after surgical resection of the tumor where tumor was removed completely with surgical specimen microscopic margins free from tumor and with available archival tumor tissue from the surgical specimen
* Patient who have AJCC 8th edition Prognostic Stage Group II
* Patient has completed adjuvant radiotherapy (if indicated) according to the institutional guidelines prior to screening
* Patient may already have initiated adjuvant endocrine therapy (ET) at the time of randomization, but randomization must take place within 52 weeks of date of initial histological diagnosis of breast cancer and within 12 weeks of initiating ET
* ECOG Performance Status 0 or 1
* Adequate bone marrow and organ function
* Sodium, potassium, phosphorus, magnesium and total calcium laboratory values within normal limits
* QTcF interval < 450 msec and mean resting heart rate 50-90 bpm

Key Exclusion Criteria:

* Prior neoadjuvant therapy (endocrine therapy or chemotherapy) or CDK4/6 inhibitor
* Prior treatment with tamoxifen, raloxifen or aromatase inhibitors for reduction in risk (chemoprevention) of breast cancer and/or treatment for osteoporosis within last 2 years
* Patient with inflammatory breast cancer
* Prior treatment with anthracyclines at cumulative doses of 450 mg/m² or more for doxorubicin or 900 mg/m² or more for epirubicin
* Distant metastases of breast cancer beyond regional lymph nodes
* Patient has not recovered from clinical and laboratory acute toxicities of chemotherapy, radiotherapy and surgery
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, or clinically significant cardiac arrhythmias
* Uncontrolled hypertension with systolic blood pressure >160 mmHg
* Patient is currently receiving any of the prohibited substances that cannot be discontinued 7 days prior to Cycle 1 Day 1: concomitant medications, herbal supplements, and/or fruits and their juices that are known as strong inhibitors or inducers of CYP3A4/5; medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5; systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment; concomitant medications with a known risk to prolong the QT interval and/or known to cause torsades de points that cannot be discontinued or replaced by safe alternative medication.
* Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the study
* Women of child-bearing potential unless they are using highly effective methods of contraception during the study treatment and for 21 days after stopping the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-31 (Estimated); Primary Completion 2025-11-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (iDFS) using STEEP criteria | up to 90 months
  iDFS is defined as the time from the date of randomization to the date of the first event of local invasive breast recurrence, regional invasive recurrence, distant recurrence, death, contralateral invasive breast cancer, or second primary non-breast invasive cancer, and is assessed locally by investigators.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) using STEEP criteria | up to 90 months
  RFS is defined as the time from date of randomization to date of first event of local invasive breast recurrence, regional invasive recurrence, distant recurrence, or death.
Distant disease-free survival (DDFS) using STEEP criteria | up to 90 months
  DDFS is defined as the time from date of randomization to date of first event of distant recurrence, death, or second primary non-breast invasive cancer
Overall survival (OS) | up to 90 months
  OS is defined as the time from date of randomization to date of death due to any cause.
Quality of Life (QOL) | Baseline, 90 months
  Change from baseline in the physical functioning sub-scale score and global health status/QOL scale score as assessed by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trials in line with applicable laws and regulations. This trial data will be available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Result] Hudis CA, Barlow WE, Costantino JP, Gray RJ, Pritchard KI, Chapman JA, Sparano JA, Hunsberger S, Enos RA, Gelber RD, Zujewski JA. Proposal for standardized definitions for efficacy end points in adjuvant breast cancer trials: the STEEP system. J Clin Oncol. 2007 May 20;25(15):2127-32. doi: 10.1200/JCO.2006.10.3523. PMID 17513820
- [Result] Hortobagyi GN, Connolly JL, D'Orsi CJ, et al (2017). Breast. From AJCC Cancer Staging Manual 8th ed. By Amin MB, Edge S, Greene FL, et al. Springer